CLINICAL TRIAL: NCT02514980
Title: Infra-orbital Nerve Block for Post Operative Analgesia in Young Children Undergoing Pediatric Cleft Lip Surgery.
Brief Title: Infra-orbital Nerve Block for Post Operative Analgesia in Children Undergoing Cleft Lip Surgery.
Acronym: IFONB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00008718/ ref. no.103
Record Dates: First submitted 2015-08-01; First posted 2015-08-04 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine group (Active Comparator): Infraorbital nerve block using bupivacaine 0.25% on each side.
  Interventions: Drug: Bupivacaine
- Bupivacaine-Ketamine group. (Active Comparator): Infraorbital nerve block using bupivacaine 0.25% combined with 0.5mg/kg ketamine on each side.
  Interventions: Drug: Bupivacaine; Drug: Ketamine

INTERVENTIONS:
Drug: Bupivacaine — Infraorbital nerve block using bupivacaine 0.25% on each side.
  Other Names: bucaine
Drug: Ketamine — Infraorbital nerve block using 0.5mg/kg ketamine on each side.
  Other Names: Katalar
  Arms: Bupivacaine-Ketamine group.

SUMMARY:
this study will be undertaken to evaluate the safety and analgesic efficacy of adding ketamine to bupivacaine in bilateral infra-orbital nerve block for relief of pain postoperatively following repair of cleft lip in children less than two years of age.

DETAILED DESCRIPTION:
Oro-facial clefts are the most prevalent craniofacial birth defects and the second most common birth anomaly, second only to clubfoot [Strong & Buckmiller 2001]. Cleft lip surgery is associated with appreciable postoperative pain in children Alleviation of postoperative pain is important in these patients. The fear of respiratory depression using opioids has renewed the interest in regional anesthesia to provide safe and effective postoperative analgesia. Infra-orbital nerve block has been advocated as a suitable local analgesic technique for cleft lip surgery and superficial surgery on the mid face [Morton 2004, Takmaz et al. 2009, Rajesh et al. 2011, Jindal et al. 2011].The infra-orbital nerve supplies the upper lip, lower eyelid, and adjacent skin of the cheek and nose. Unilateral or bilateral infra-orbital nerve block has been performed with a very high success rate.

The investigators designed this study to evaluate the safety and analgesic efficacy of adding ketamine to bupivacaine in bilateral infra-orbital nerve block for relief of pain postoperatively following repair of cleft lip in children less than two years of age.

ELIGIBILITY:
Inclusion Criteria:

(ASA) physical status I and II aged less than 2 years undergoing elective cleft lip repair (with or without cleft palate) under general anesthesia.

Exclusion Criteria:

Patients with local infection at the site of injection of block, history suggestive of drug allergy, any systemic disease that compromises the cardiovascular, respiratory or neurological function, other congenital anomaly, history of upper or lower airway disease, coagulation disorders, and children with history of sleep apnea and in whom postoperative ventilation may be required will be excluded from the study.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
postoperative analgesic consumption | 24 hours postoperative
  the total consumption of analgesics in the first 24h postoperative

SECONDARY OUTCOMES:
Postoperative The Face, Legs, Activity, Cry, Consolability ( FLACC) pain score | 24 h postoperative.
  FLACC pain score will be recorded on arrival to the recovery room (0) and at 1, 2, 3, 4, 8, 12, and 24 hours postoperative.
Parent satisfaction score | 24 h postoperative
  The parents will be asked to evaluate their satisfaction regarding pain control at the end of 24 hours over a score of 4 points (1=bad, 2=moderate, 3=good, 4=excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in Anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
This is a single center study with no plan to share data